## A Research Inquiry: Examining Engagement Trends Among Participants in Hidradenitis Suppurativa Clinical Trials

An Informed Consent Form For <u>Power Clinical Trial's</u> Hidradenitis Suppurativa Observational Clinical Study

Date: December 29, 2023

Introduction to the Informed Consent Form: A Brief Overview

This summary serves to outline our observational clinical study, highlighting its procedures, potential risks, and participant benefits. While your consent is necessary, your involvement is voluntary, granting you the freedom to withdraw without repercussions.

Our study aims to grasp the reasons behind hidradenitis suppurativa patients' choices to engage, persist, or discontinue participation in clinical trials. The primary processes include questionnaire completion and follow-up calls, designed to mitigate participant risks.

Although direct medical benefits may not accrue to participants in this observational study, the compiled data will aid in identifying methods to enhance clinical trial participation rates, ultimately benefiting individuals with hidradenitis suppurativa.

The study's conclusions will yield crucial insights into the factors impacting clinical trial participation rates. Our goal is to refine recruitment approaches and bolster patient involvement in trials, leading to improved treatment options and outcomes for hidradenitis suppurativa sufferers. However, engaging in this study is voluntary, and declining will not affect your rights.

Carefully reviewing the consent form and seeking clarification on any concerns is paramount before reaching a decision. It's advisable to engage in discussions with family, friends, advisors, and healthcare professionals to ensure a well-informed choice.

Engagement remains completely optional, allowing withdrawal at any point without repercussions.

Analyzing Engagement Determinants in Hidradenitis Suppurativa Clinical Studies

Clinical trials play a pivotal role in advancing hidradenitis suppurativa treatments, yet concerns persist about the representativeness of trial participants. This study aims to uncover the factors driving patient decisions regarding enrollment, withdrawal, or re-engagement in hidradenitis suppurativa clinical trials. Understanding these factors will significantly improve the relevance and effectiveness of future research endeavors.

To ensure comprehensive insights, our focus is on recruiting a diverse demographic spectrum. Investigating how variables like age, race, income, and education influence participation decisions is critical. This collected data aims to develop more effective strategies for engaging underrepresented groups in forthcoming clinical trials.

Participation in this study is entirely voluntary, allowing individuals to withdraw at any point without facing consequences. The study procedures, involving questionnaire completion and follow-up calls, pose minimal risks to participants. Prospective participants are strongly encouraged to meticulously review the consent form and seek clarification for any queries.

Ultimately, this trial endeavors to deepen our understanding of the factors impacting hidradenitis suppurativa clinical trial participation. Enhancing participation rates could accelerate the development of innovative treatments for this debilitating condition.

Investigating Engagement in Hidradenitis Suppurativa Clinical Trials

Our research delves into understanding the key drivers impacting the decisions of hidradenitis suppurativa patients regarding their participation in clinical trials. We aim to identify potential participants from past or ongoing interventional trials by utilizing electronic medical records.

Upon expressing interest, participants will receive a comprehensive consent form detailing the study's objectives and their rights. The data collection process will involve biweekly questionnaires covering demographics, medical history, and motivations guiding their involvement. Furthermore, we plan to conduct in-depth quarterly phone or video interviews for a more comprehensive understanding.

The statistical analysis of the amassed data aims to reveal the myriad of factors shaping patient involvement in clinical trials. Disseminating these findings through conferences and academic publications aims to benefit all stakeholders within clinical trial spheres.

Our goal is to leverage these discoveries to refine and strengthen future clinical studies for hidradenitis suppurativa patients, enhancing both recruitment strategies and retention rates.

Participation in this study is entirely voluntary, ensuring withdrawal at any point without any repercussions. The potential risks involve completing questionnaires and participating in follow-up interviews. Any questions or concerns can be addressed promptly by our accessible research team.

Assessing Risks in Observational Studies of Hidradenitis Suppurativa

In observational clinical research studies focused on hidradenitis suppurativa, there are no experimental treatments involved, yet participation might carry potential risks. These risks could include breaches of privacy, emotional distress related to the study's subject matter, and possible adverse outcomes from trial-associated procedures.

Before deciding to participate, it is essential to carefully examine and comprehend the informed consent form and raise any concerns with the research team. The team will offer comprehensive insights into potential risks, the benefits of the study, and safety measures in place to protect participants' welfare.

Grasping the Potential Advantages of Hidradenitis Suppurativa Observational Trials

Engaging in observational clinical trials dedicated to hidradenitis suppurativa provides patients with an opportunity to contribute to medical progress and potentially improve

forthcoming treatment options. Even without experimental therapies, patients can receive attentive care throughout the study duration.

Before committing to trial participation, patients should carefully evaluate potential benefits and risks, considering their unique circumstances and objectives. Seeking advice from healthcare providers and the research team is imperative to make a well-informed decision.

## Pondering Factors Influencing Your Decision to Participate

Recognizing that your engagement in a clinical trial might be stopped without your explicit agreement is essential. There are various reasons why researchers or sponsors may halt the trial, including study suspension, withdrawal of funding, or if it's deemed advantageous for your well-being.

Additionally, your participation may conclude due to health deterioration, pregnancy, opting out following significant updates, or failure to comply with study protocols. Thoughtfully considering these factors before embarking on a clinical trial is paramount.

Understanding Atopic Dermatitis Trials: A Comparative Outlook

Participation in atopic dermatitis clinical trials is entirely elective, ensuring individuals the liberty to withdraw without encountering adverse effects.

For a broad perspective on <u>hidradenitis suppurativa research</u> globally, clinicaltrials.gov, managed by the National Institutes of Health (NIH), stands as a comprehensive repository of trials. Users have the ability to customize their search based on geographic location and particular medical conditions.

Moreover, Power's reference page offers an updated roster of active <u>hidradenitis</u> <u>suppurativa clinical trials</u> currently open for enrollment.

Exploring Diversity in Clinical Trials Through Online Resources

Various online platforms cater to those interested in comprehending the intricacies of clinical trial diversity. Below are a couple of articles that may capture your interest:

Farb, Andrew, Charles J. Viviano, and Michelle E. Tarver. "Diversity in Clinical Trial Enrollment and Reporting—Where We Are and the Road Ahead." *JAMA cardiology* 8, no. 9 (2023): 803-805.

Gray, Darrell M., Timiya S. Nolan, John Gregory, and Joshua J. Joseph. "Diversity in clinical trials: an opportunity and imperative for community engagement." *The Lancet Gastroenterology & Hepatology* 6, no. 8 (2021): 605-607.

These resources provide insightful information regarding the challenges associated with clinical trial diversity and potential solutions.

## Safeguarding Privacy in Research Investigations

Preserving the confidentiality of the data collected in this research stands as our paramount concern. While absolute confidentiality can't be assured universally, stringent measures are in place to safeguard it. Be aware that legal requirements might demand the disclosure of personal information. Nonetheless, any research publications or presentations will refrain from disclosing your name or personally identifying details.

Various entities, such as accrediting bodies, government regulatory authorities (like the FDA and OHRP), safety monitors, study sponsors, and authorized representatives, may access your medical information for purposes related to research, quality assurance, and data analysis.

In rare instances, we may require an "Authorization Form" outlining the utilization and sharing of your information for this study. Prior to sharing your information or research samples with Power researchers, other university establishments, or external commercial entities for prospective research, explicit consent will be sought. Your confidential data will be handled securely and deleted.

## **Consent Agreement Understanding**

By signing this consent agreement, you confirm your understanding and acceptance of the following:

- Thoroughly comprehending and grasping the contents of this informed consent form, with encouragement to seek additional viewpoints before reaching a decision.
- Satisfaction with the responses provided to all your inquiries regarding the research project and its methodologies, ensuring you possess the essential information for study participation.
- Deliberation on potential benefits, drawbacks, and alternatives linked to involvement in the research.
- Acknowledgment that your voluntary participation in the research study won't impede your legal rights.
- Assurance of timely communication regarding any significant updates that might influence your decision to continue participating in the research study.
- Provision of this consent form, affording you the opportunity to address any lingering questions.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Affirmation by the Investigator | | |
| In my capacity as the investigator, I haddressed, fostering a comprehensive reaffirmed that the patient's participat | e understanding of the study. | Moreover, I have |
| Signature of Researcher Who R | Received Consent | |
| Name of Investigator | Signature of Investigator | Date |